CLINICAL TRIAL: NCT05073354
Title: Implementation of a Mobile In-hospital Resuscitation Model for the Rapid Treatment of Shock Without Trauma (SWOT)
Brief Title: Rapid Treatment of Shock Without Trauma
Acronym: SWOT
Status: Completed | Type: Observational
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 50701
Record Dates: First submitted 2021-09-28; First posted 2021-10-11 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Shock
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Full-implementation: Patients experiencing shock without trauma once all training is in place and devices are deployed
  Interventions: Device: Full SWOT Model

INTERVENTIONS:
Device: Full SWOT Model — Bundle of care that includes devices such as X Series monitor/defibrillator, AutoPusle automated compression device, Z Vent ventilator, and IPR therapies as well as bedside monitoring and diagnostics and training on a standardized care process.

SUMMARY:
Evaluate the implementation of a standardized mobile resuscitation model to manage SWOT within a large acute care hospital setting.

DETAILED DESCRIPTION:
Immediately upon identification of SWOT, the SWOT Team will be activated by clinicians to respond to the patient bedside. Clinicians on-site will initiate patient care as directed by hospital protocol. Upon arrival, the SWOT Team will take over the management of patient care. The team will include 1-2 intensivists and multiple clinicians with clearly defined roles, dependent upon clinical presentation. The mobile resuscitative platform equipped with critical care technology will be delivered to the bedside (refer to appendix for full equipment content).

The SWOT Team will implement goal-directed therapy using real-time monitoring and advanced diagnostic point-of-care tools. ultrasound, arterial and central lines will be placed by the intensivist(s) to monitor the physiology of the patient during treatment in real-time. Other team members (RNs, Respiratory Therapist's, residents, anesthesiologists, and technicians) will place the patient on continuous ECG and SPO2 monitoring, continuous capnographic monitoring via nasal canula or Endotracheal tube, and continuous cerebral and regional NIRS monitors. Point-of-care laboratory values will also be measured. Resuscitative interventions will be performed as directed by team leader to target the following physiological target parameters:

* SpO2 > 85%
* PaO2 > 50 mmHg
* NIRS > 65%
* Lactate normal or trending down
* EtCO2 >20 mmHg
* Mean Arterial Pressure > 65 mmHg
* SVO2 > 60%

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years of age (inclusive)
2. Presence of shock, defined as systolic blood pressure (SBP) less than 90 mmHg with signs of hypoperfusion, including at least one of the following (without alternate causes):

   * low cardiac index (<2.2 L/min/m2)
   * elevated filling pressures of the left heart (pulmonary capillary wedge pressure [PCWP] >15 mmHg) and/or
   * right heart (central venous pressure [CVP] >10 mmHg)
   * non-perfusing cardiac rhythm or cardiac arrest
   * mixed venous oxygen saturation <60% or >80% without non-shock cause
   * Heart rate >90 beats per minute
   * Respiratory rate >20 breaths per minute
   * White blood cell count >12 or < 4
   * Temperature >38°C or <35°C
   * SOFA score ≥2 with vasopressor requirement and elevated lactate >2 mmol/L (>18 mg/dL) despite adequate fluid resuscitation
   * Central venous pressure <8 mmHg
   * Obstruction such as pulmonary embolus on imaging
3. Admitted to Abbott Northwestern
4. Rapid Response Team call or request
5. Patients who previously agreed to allow their medical record information to be used for Allina Health research (i.e. Minnesota Research Authorization (MRA) "Yes") or those who have not explicitly declined use of their medical information in Allina Health research (i.e. MRA "Null")

Candidates for the prospective case series must meet the following inclusion criterion:

1. Interventional assessment and treatment by SWOT Team (full-implementation period only)
2. Patients who previously agreed to allow their medical record information to be used for Allina Health research (i.e. Minnesota Research Authorization (MRA) "Yes") or those who have not explicitly declined use of their medical information in Allina Health research (i.e. MRA "Null")

Exclusion Criteria:

1. Known or suspected pregnancy
2. Significant trauma
3. BMI > 50 kg/m2
4. Pre-existing Do Not Resuscitate order
5. Presence of orders limiting resuscitation efforts during the initial resuscitative period (less than 2 hours from the onset of protocol)
6. Refusal to receive whole blood or blood products
7. Severe brain injury (anoxic, traumatic, hemorrhagic or ischemic)
8. presence of an assist device such as intra-aortic balloon pump
9. Advanced chronic organ dysfunction
10. Known or presumed COVID-19
11. Patients with a status of MRA "No"
12. Patient in ICU at time of shock

Candidates for the prospective case series will be excluded if the following condition is present:

1. Patients with a status of MRA "No"
2. Patient in ICU at time of shock

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients meeting all enrollment criteria will be eligible for enrollment in the study.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Time to Shock Reversal | From 24 hours to 72 hours after initial shock event
  Duration in minutes from activation of the SWOT Team to shock reversal, defined as stable arterial pressure (SBP > 90 mmHg) without requirement for vasopressor administration for greater than 24 hours and normalization of systemic and local perfusion measures of lab-measured lactate indicating improved systemic perfusion

SECONDARY OUTCOMES:
30-day Mortality | 30 days after initial shock event
  Patient all-cause mortality will be assessed at 30 days following initial identification of shock symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Tonia M Mowbray-Donahue, MD, Principal Investigator — Allina Health
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No